CLINICAL TRIAL: NCT04521465
Title: A Multi-Center, Single Arm, Post-Market Clinical Follow-up Study to Evaluate the Safety and Efficacy of NovaTears® + Omega-3 (0.2%) Eye Drops on Signs and Symptoms of Dry Eye
Brief Title: Safety and Efficacy of NovaTears® + Omega-3 (0.2%) Eye Drops on Signs and Symptoms of Dry Eye
Status: Completed | Type: Observational
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NTO-001
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Evaporative Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NovaTears® + Omega-3
  Interventions: Device: NovaTears® + Omega-3 (Perfluorohexyloctane with 0.2% w/w Omega-3 fatty acid ethyl esters)

INTERVENTIONS:
Device: NovaTears® + Omega-3 (Perfluorohexyloctane with 0.2% w/w Omega-3 fatty acid ethyl esters) — Eye drops

SUMMARY:
This PMCF study is carried out following successful CE marking of NovaTears® + Omega-3 and is intended to generate systematic clinical data on the safety and performance of the device when used in accordance with the intended purpose.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form) and data protection form
* Patient-reported history of DED in both eyes
* Have an Ocular Surface Disease Index (OSD) score ≥ 25 at Visit 1
* Have Meibomian Gland Dysfunction (MGD) at Visit 1.
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning a pregnancy
* Ocular surface pathology, clinically significant slit-lamp findings, abnormal lid anatomy, active ocular allergies
* Wear of contact lenses
* Known allergy or sensitivity to the medical device or its components
* Currently enrolled in an investigational drug or device study or have used an investigational drug or device within 60 days before Visit 1.
* Clinical site employees or immediate family members of the same

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with evaporative Dry Eye Disease
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to confirm the performance, relieving symptoms and improving signs of DED, and to evaluate safety and tolerability of topical NovaTears® + Omega-3 (0.2%) eye drops, when used in accordance with its approved labeling | 2 months
  This PMCF study is intended to provide systematic clinical data supporting the safety and performance of the medical device NovaTears® + Omega-3 (0.2%).

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH
Locations (2):
- Germany (2):
  - NTO-001 Investigational Site, Heidelberg
  - NTO-001 Investigational Site, Nuremberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobi C, Angstmann-Mehr S, Lange A, Kaercher T. A Water-Free Omega-3 Fatty Acid Eye Drop Formulation for the Treatment of Evaporative Dry Eye Disease: A Prospective, Multicenter Noninterventional Study. J Ocul Pharmacol Ther. 2022 Jun;38(5):348-353. doi: 10.1089/jop.2021.0102. Epub 2022 May 4. PMID 35507946